CLINICAL TRIAL: NCT03431948
Title: Platform Phase 1 Study Investigating the Safety of Stereotactic Body Radiotherapy (SBRT) With Immuno-oncology Agents for the Treatment of Multiple Metastases in Advanced Solid Tumors
Brief Title: Stereotactic Body Radiotherapy (SBRT) Plus Immunotherapy for Cancer
Acronym: C4-MOSART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-1317; CA025-002 (Other: Bristol Myers Squib)
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; cabiralizumab; urelumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled in parallel based on physician preference and slot availability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SBRT with Nivolumab and Urelumab (Experimental): Patients will receive stereotactic body radiation therapy (SBRT) in combination with nivolumab and urelumab.
  Interventions: Drug: Nivolumab; Drug: Urelumab; Radiation: Stereotactic Body Radiation Therapy
- SBRT with Nivolumab and Cabiralizumab (Experimental): Patients will receive stereotactic body radiation therapy (SBRT) in combination with nivolumab and cabiralizumab .
  Interventions: Drug: Nivolumab; Drug: Cabiralizumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240 mg given by intravenous infusion every 2 weeks
  Other Names: OPDIVO; BMS-936558
Drug: Cabiralizumab — Cabiralizumab 4 mg/kg given by intravenous infusion every 2 weeks
  Other Names: BMS-986227; FPA008
  Arms: SBRT with Nivolumab and Cabiralizumab
Drug: Urelumab — Urelumab 8 mg given by intravenous infusion every 4 weeks
  Other Names: BMS-663513
  Arms: SBRT with Nivolumab and Urelumab
Radiation: Stereotactic Body Radiation Therapy — Radiation to metastatic lesion(s) given at assigned dose levels based on lesion location and dose level being tested at time of enrollment. Doses range from 30 - 50 Gy.

SUMMARY:
Study to determine the best dose of stereotactic body radiation therapy (SBRT) to be administered in combination with immunotherapy drugs including urelumab, cabiralizumab and nivolumab .

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide written informed consent
* Willingness and ability to comply with required study visits and procedures
* For Biopsy Patients: Willingness to undergo repeat biopsy of tumor before and after treatment
* Men or women ≥ 18 years of age.
* Histologically confirmed advanced solid tumor for which curative treatment is not available.
* Have undergone appropriate standard of care treatment options (in the opinion of the treating investigator). Participants with NSCLC must have undergone EGFR and ALK testing and have received appropriate initial therapy.
* Measurable disease, including at least one tumor lesion that meets criteria for multi-organ site ablative radiation therapy (MOSART) SBRT radiation.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Adequate organ function, as defined by the following:
* Absolute neutrophil count (ANC) ≥ 1,500/µL
* Platelets ≥ 100 x 10^3/µL
* Hemoglobin ≥ 8 g/dL without transfusion or EPO dependency
* Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCL) > 50 mL/min (creatinine clearance should be calculated per institutional standard). GFR can also be used in place of creatinine of CrCl.
* Serum total bilirubin ≤1.5 x institutional ULN (except subjects with Gilbert's Syndrome, who must have normal direct bilirubin).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x institutional ULN OR ≤ 5x ULN for subjects with liver metastases.
* Albumin > 3.2 mg/dL.
* Prior immuno-oncology (IO) therapy
* Have a physician determined life expectancy of at least 6 months.
* Negative pregnancy test for women of childbearing potential (WOCBP) within 72 hours of starting therapy
* Must not be breastfeeding
* Woman of childbearing potential: Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) and up to 5 months post last dose of study drug(s).
* Men: Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) and up to 7 months post last dose of study drug(s). Must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Must not be currently receiving study therapy or have participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Must not have had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or have not recovered (i.e. < grade 1 at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Must not have had prior chemotherapy, targeted small molecule therapy, radiation or other anti-cancer therapy (with exceptions for disease-specific hormone treatments considered standard of care) within 2 weeks prior to study Day 1 or have not recovered (i.e. < grade 1 or at baseline) from adverse events due to a previously administered agent. Exception for ≤ grade 2 neuropathy. If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Must not have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable, have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Must not have had prior radiation therapy (defined as >10% of prior prescription dose) to the area planning to be treated with SBRT.
* Must not have a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a dose of >10 mg prednisone daily or equivalent at time of first dose of trial treatment.
* Must not have a known history of active TB (Bacillus Tuberculosis)
* Must not have hypersensitivity to nivolumab, urelumab, cabiralizumab or any of their excipients.
* Must not have a known additional malignancy that could confuse analysis of on-study treatment. Inclusion of all study participants with more than one malignancy must be discussed and approved by the PI.
* Must not have active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroids replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Must not have a known history of non-infectious pneumonitis that required steroids for treatment.
* Must not have evidence of interstitial lung disease.
* Must not have an active infection requiring systemic therapy.
* Must not have a history or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* If known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) then patient is not eligible for cohorts including SBRT to liver lesions.
* Participants must not have had prior organ allograft or allogeneic bone marrow transplantation.
* Participants must not have had uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction or stroke/transient ischemic attack within the past 6 months
  * Uncontrolled angina within the past 3 months
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  * History of other clinically significant heart disease (eg, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, significant pericardial effusion, or myocarditis)
  * Cardiovascular disease-related requirement for daily supplemental oxygen therapy
* Has received a live vaccine within 30 days of planned start of study therapy.
* Participants may not concomitantly use statins while on study. However, a patient using statins for over 3 months prior to study drug administration and in stable status without CK rise may be permitted to enroll.
* Participants may not have current or history of clinically significant muscle disorders (eg, myositis), recent unresolved muscle injury, or any condition known to elevate serum CK levels.
* Must not have a history of allergy to nivolumab, urelumab or cabiralizumab.
* Must not have a history of any significant drug allergy (such as anaphylaxis or hepatotoxicity) to prior anti-cancer immune-modulating therapies (eg, checkpoint inhibitors and T-cell co-stimulatory antibodies).
* Must not be prisoners or be involuntarily incarcerated.
* Must not be compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Recommended dose of SBRT given in combination with immunotherapy | 3 months
  Dose of stereotactic body radiation therapy (SBRT) that can safety be given with immunotherapy.

SECONDARY OUTCOMES:
Rates of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher side effects | 3 months
  Rate of side effects seen in study participants.
Rates of long term side effects | 6 - 24 months
  Rate of long term (occurring 6 month or more after treatment) side effects seen in study participants.
Response rate | 6 months
  Rates of response (tumor shrinkage).
Progression free survival rate | 6 months
  Number of participants that do not have disease worsening.
Overall survival rate | 6 - 24 months
  Number of participants still alive.
Local disease control of SBRT treated lesions | 6 months
  Rate of disease control (tumor shrinkage) of radiation treated lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Luke, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided